CLINICAL TRIAL: NCT04237220
Title: Comparison of Two Methods for Endoscopic Biopsy to Detect Helicobacter Pylori
Brief Title: Endoscopic Biopsy to Detect Helicobacter Pylori
Status: Completed | Type: Observational
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, Dr. med. Hector Eloy Tamez Perez, Clinical professor, Hospital Universitario Dr. Jose E. Gonzalez
Other Study IDs: GA19-00004
Record Dates: First submitted 2020-01-17; First posted 2020-01-23 (Actual); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: Helicobacter Pylori Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Stomach biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: stomach biopsies — To determine the diagnostic performance in the detection of Helicobacter pylori in biopsies taken only from the gastric antrum for the determination of the positive predictive value, the negative predictive value, and sensitivity and specificity.

SUMMARY:
Helicobacter pylori (H. pylori) infection represents one of the most common chronic infections that affect humans.Endoscopy must be performed to take biopsies for detection of Helicobacter pylori in patients with alarm symptoms. The Sydney Protocol is the recommended strategy that guarantees maximum diagnostic yield. This is a prospective uncontrolled cross-sectional clinical trial.

Endoscopy must be performed to take biopsies for detection of Helicobacter pylori in patients with epigastric pain, weight loss, iron-deficiency anemia, individuals with dyspepsia over 60 years of age or younger with alarm symptoms (weight loss, dysphagia, vomiting, gastrointestinal bleeding, among others).

The Sydney Protocol is the recommended strategy that guarantees maximum diagnostic yield. Histology is expensive since it requires time for biopsy processing and trained personnel for staining and interpretation but it provides additional information on the degree of inflammation and complications such as atrophic gastritis, intestinal metaplasia, and malignancy. The modified Sydney protocol includes two biopsies from the antrum, two from the body, and one form the incisura.

DETAILED DESCRIPTION:
The hypothesis is that the histopathological study of two biopsies obtained from the gastric antrum for the determination of Helicobacter pylori infection has a similar diagnostic yield compared to the gold standard (Sydney protocol). This is a prospective uncontrolled cross-sectional clinical trial.

Patients older than 18 years with a medical indication for performing upper gastrointestinal endoscopy for biopsy and detection of Helicobacter pylori infection in the period from january to May 2020.

A sample size of 67 patients was calculated using the diagnostic test comparison formula, in order to compare the sensitivity and specificity in patients with indications for a biopsy taken with the Sydney protocol from those taken only from the gastric antrum.

Expecting a sensitivity of 89% in the Sydney protocol With a Zα of 1.96 and a maximum amplitude of 7.5% (CI = 15), at least 67 study subjects are required with the two diagnostic tests.

Cold biopsies will be taken using an oval head clamp with a stiletto, 2.3 mm in diameter and 180 cm in length of the gastric mucosa with the current standardized method (Sydney protocol).

The samples will be sent to the pathology service in two bottles with formalin; in one, the two biopsies obtained from the antrum will be labeled as "bottle 1" and in the second bottle obtained from the body and the incisura will be labeled as "bottle 2"; this will be blinded for the pathologist who analyzes the slides.

Samples will be processed in a conventional manner, stained for interpretation with hematoxylin-eosin and Giemsa.

Upon obtaining the pathology report, the data will be analyzed in the SPSS statistical program by 2X2 contingency tables for the determination of the positive predictive value, the negative predictive value, and the sensitivity and specificity of the biopsies taken from the antrum compared to healthy population and those who possess the infection using the gold standard.

In addition, the diagnostic yield of the biopsies taken from the antrum of patients who use PPI or have atrophic gastritis will be analyzed separately.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years
* Have a clinical file.
* Medical indication for upper gastrointestinal endoscopy and biopsy to detect Helicobacter pylori

Exclusion Criteria:

* Active gastrointestinal bleeding
* Antibiotic use in the last 30 days
* Hemodynamic instability
* Platelets <50,000 K/µL
* INR >1.5 or PT >50 sec
* Having received eradication treatment for Helicobacter pylori previously.
* History of gastric surgery
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients attending the outpatient Gastroenterology clinic and the Emergency Department of the "Dr. Jose Eleuterio González" University Hospital with a medical indication for performing upper gastrointestinal endoscopy for biopsy and detection of Helicobacter pylori infection.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2020-01-25 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-05-20 (Actual)

PRIMARY OUTCOMES:
2 Antrum biopsy diagnostic performance | 7 days
  To determine the diagnostic performance in the detection of Helicobacter pylori in biopsies taken only from the gastric antrum for the determination of the positive predictive value, the negative predictive value, and sensitivity and specificity.

CONTACTS AND LOCATIONS:
Overall Officials: Joel O. Jáquez, M.D., Study Director — Hospital Universitario
Locations (1):
- Hospital Universitario Dr. Jose E. Gonzalez, Universidad Autónoma de Nuevo León, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No